CLINICAL TRIAL: NCT02995850
Title: A Phase Ib/II Study of Efficacy and Feasibility of Cytoreductive Surgery, Extensive Peritoneal Lavage, Hyperthermicintraperitoneal Chemotherapy and Post-operative Intraperitoneal Chemotherapy Combination in Gastric Cancer With Peritoneal Metastasis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 4-2016-0252
Record Dates: First submitted 2016-12-14; First posted 2016-12-19 (Estimated); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Gastric Cancer With Peritoneal Metastasis (PCI<12)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anti-cancer drug (Experimental)
  Interventions: Drug: CRS+HIPEC

INTERVENTIONS:
Drug: CRS+HIPEC — 1. Ib
     * Dose-escalation of intraperitoneal paclitaxel will follow a modified 3 + 3 dose escalation procedure.
  2. II
     ① CRS If PCI <12, CRS will be performed by gastrectomy with D2-lymphadenectomy and resection of any involved adjacent structures.
     If PCI≥12, instead of CRS, 3 times of IP paclitaxel +cisplatin and oral S-1 chemotherapy every 3 weeks, and then PCI <12, CRS will be done.
     ② Extensiveintraperitoneal lavage Peritoneal lavage after CRS will be done with 10 L before HIPEC.
     ③ HIPEC Following surgery HIPEC will be performed using CDDP (60 mg/m2) and PTX (P2RD mg/m2). IP chemotherapy will be performed.
     ④ Post-operative intraperitoneal chemotherapy Postoperative chemotherapy will be done 8 cycles of IP paclitaxel+ cisplatin and oral S-1 after 4 weeks.

SUMMARY:
This is an open-label, non-randomized, single-center, phase Ib/II study, evaluating efficacy and feasibility of cytoreductive surgery(CRS), extensive peritoneal lavage, hyperthermic intraperitoneal chemotherapy(HIPEC) and post-operative intraperitoneal chemotherapy combination in gastric cancer with peritoneal metastasis

DETAILED DESCRIPTION:
Peritoneal metastases in gastric cancer are considered to indicate terminal disease due to poor prognosis because systemic chemotherapy is unlikely to accumulate in peritoneal nodules in cytotoxic concentrations. Cytoreductive surgery (CRS) along with hyperthermic intraperitoneal chemotherapy (HIPEC) has been suggested to improve survival in select patients with limited peritoneal spread, resulting in a median overall survival (OS) of 8 to 14 months. It remains unclear, however, which regimen is best and who have benefits from CRS and HIPEC. Herein, we has conducting prospective phase Ib/II trial of CRC and HIPEC with intraperitoneal paclitaxel and cisplatin, and oral S-1 in gastric cancer with peritoneal metastasis.

ELIGIBILITY:
Inclusion Criteria:

1. Patient age of 19 years or older and age of 75 years or younger.
2. Histologically proven gastric or esophagogastric junction adenocarcinoma with peritoneal metastasis under diagnostic laparoscopy.
3. Primary tumor measured as resectable in preoperative images.
4. Performance status based on ECOG : 0~1
5. No prior treatment (chemotherapy, radiotherapy, etc.)
6. Adequate hepatic, renal, and hematologic function

   * ANC≥1,500/uL,
   * hemoglobin≥9.0g/dL
   * platelet≥100,000/uL
   * total Bilirubin: ≤ 1.5 × upper normal limit
   * Creatinine<1.5mg/dL
   * AST/ALT, ALP ≤ 2.5 x upper normal limit
7. Patients who can understand this study and sign the consent form.

Exclusion Criteria:

1. Patient who has distant metastasis or para-aortic lymph node metastasis or retroperitoneal metastasis except peritoneal metastasis. (But the patient who has ovarian metastasis with resectable status can be enrolled.)
2. Primary tumor cannot be resected because of direct invasion to other important organ. (But, if the invaded organ can be resected together, such as spleen, gallbladder, distal pancreas, and liver, the patient can be enrolled)
3. HER2 positive patient
4. Patient with active viral infection (for example, HIV, HBV, HCV, except stable status of HBV infection)
5. Pregnant patient, or patient in breast-feeding, or who is planning pregnancy.
6. Patients in exclusion criteria of TS-1, cisplatin, paclitaxel

   * Patients with a history of severe hypersensitivity to these drugs
   * Patients with severe bone marrow depression
   * patients who has severe hepatic, renal disorder
   * patients who has hereditary problem or galactose intolerance, lapp lactase deficiency, or glucose-galactose malabsorption
7. Patients who has important medical problem or infection

   * Cerebrovascular accident(CVA) within 1 year
   * Heart attack within 6 months, uncontrolled hypertension, unstable angina, uncontrolled congestive heart failure(CHF), severe arrhythmia
   * Major operation or injury within 28 days
   * Severe and not recovered wound, ulcer, fracture
   * Uncontrolled bleeding disease
   * Recent active gastric infection
8. Patient with another primary cancer within last 5 years
9. Patient on medication which can interact with the drugs used in this study (fluoropyrimidine-group antineoplastic agents, flucytosine, phenytoin, etc)
10. Patients with other systemic chemotherapy or radiotherapy
11. Patients with psychiatric or neurologic disorder so that he or she cannot understand and sign the consent form.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-02-22 (Actual); Primary Completion 2022-04-19 (Actual); Study Completion 2022-05-05 (Actual)

PRIMARY OUTCOMES:
Ib: Maximum tolerate dose | 3 months
  Ib: To determine the MTD of orally administered S-1 + intraperitoneal paclitaxel +cisplatin in gastric cancer with peritoneal metastasis.
II: Safety | 3 months
  II:To assess the safety and tolerability of CRS +HIPEC (Clavien-Dindo classification of surgical complication & NCI-common terminology criteria for adverse events(CTC-AE) for chemotherapy]

SECONDARY OUTCOMES:
OS (overall survival) | 12 months
  the length of time from the patient signing the consent form until the patient is still alive
PFS (Progression-free survival) | 12 months
  the length of time from the patient signing the consent form until the patient shows disease progression
RR (response rate) | 12 months
  the proportion of complete response to partial response These will be estimated by the Kaplan-Meire method.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Surgery, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided